CLINICAL TRIAL: NCT02086318
Title: A New Algorithm to Predict Ovarian Age Combining Clinical, Biochemical and 3D-ultrasonographic Parameters: OvAge
Brief Title: A New Algorithm to Predict Ovarian Age
Acronym: OvAge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Other Study IDs: OvAge
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Infertility; Polycystic Ovary Syndrome; Premature Ovarian Failure (POF); Ovarian Cysts; Endometriosis
Keywords: Ovarian reserve; Ovarian age; Fertility; Reproductive prognosis; Distance to menopause
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome; Primary Ovarian Insufficiency; Ovarian Cysts; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OvAge assessment: Basal serum anti-Mullerian hormone (AMH), Follicle-stimulating hormone (FSH) and estradiol (E2), antral follicle count (AFC), ovarian volume, Vascularization Index (VI), Flow Index (FI) and Vascularization Flow Index (VFI) will be measured in all women between day 1 and day 4 of menstrual cycle
  Interventions: Other: OvAge assessment

INTERVENTIONS:
Other: OvAge assessment — Basal serum anti-Mullerian hormone (AMH), Follicle-stimulating hormone (FSH) and Estradiol (E2), antral follicle count (AFC), ovarian volume, Vascularization Index (VI), Flow Index (FI) and Vascularization Flow Index (VFI) will be measured in all women between day 1 and day 4 of menstrual cycle. Evaluation can be repeated after every kind of intervention regarding ovaries, both medical or surgical. Evaluation can be repeated also at interval of 3-6-12 months in order to study the modification of ovarian age when time passes.

SUMMARY:
To collect data of clinical, biochemical and 3D-ultrasonographic parameters of a population of fertile women aged 18-55 in order to design a new algorithm able to predict ovarian age and to evaluate the reliability of a multimodal diagnostic evaluation of ovarian age in term of both reproductive prognosis and distance to menopause following the guidelines of the Standards for Reporting of Diagnostic Accuracy initiative (STARD)

DETAILED DESCRIPTION:
The normal process of reproductive aging varies considerably among women. This implies that some women remain highly fertile until the fifth decade of their life, whereas others face the loss of natural fertility already in their mid-thirties. Female reproductive aging seems to be largely based on age related changes in ovarian function. Decreasing numbers of follicles, coinciding with diminished oocyte quality, dictate the gradual changes in menstrual cycle regularity and monthly fecundity which inevitable evolution will be menopause. The mechanisms behind the observed gradual decline of the follicle pool and the reduced oocyte quality are far from being fully understood, although recent knowledge regarding the endocrine, paracrine, genetic, and metabolic factors involved has led to a better understanding of this immensely complex puzzle.

Within the context of normal female reproductive aging, as already outlined, large individual variation exists in the age at which the various reproductive events occur. This variation has major implications for the preventive management of age-related decreased fertility and general health risks associated with extremely early menopause in conditions such as POF. Moreover, distance from menopause is an important parameter which can lead clinician's choice in the appropriate timing for surgical treatment of benign gynecological pathologies.

Although chronological age is the most important predictor of physiological ovarian response to endogenous and exogenous Follicle-stimulating Hormone (FSH), both environmental and genetic factors contribute to biological ovarian ageing, so that chronological and biological age are not always equivalent. Among genetic factors able to determine age at which menopause will occur, the most important are the size of the initial oocyte stock, the proportion that undergoes atresia and the rate of initiation of follicles growth. It has been suggested, moreover, that certain single nucleotide polymorphisms (such as regarding FSH receptors genotype) also affect sensitivity to gonadotrophins and ovarian ageing [Alviggi 45]. Environmental factors such as diet, cigarette smoking, regimens of chemotherapy or radiotherapy, endometriosis or ovarian surgery may shorten the functional lifespan of a woman's ovaries too.

Even if the continuous follicles loss will only be recognized in the late stages by cycle irregularity, endocrine and ultrasound markers have emerged over the last decade that may express more accurately the follicle number decline over a long time period. Among endocrine parameters, the most studied and used in clinical practice are FSH, Estradiol (E2) and Anti-Mullerian Hormone (AMH).

Basal FSH, extensively studied over the past few decades, provides the most indirect marker of ovarian reserve. FSH levels increase with advancing age, by reducing the negative feedback on FSH release from the pituitary [broekm vecchio 10]. High FSH levels therefore represent small cohort size. To exclude the possibility that confounding factors, such as E2 levels greater than 50 pg/ml, suppress FSH secretion, this parameters have to be always evaluated together on menstrual cycle days 1-4.

In women with varying degrees of hypergonadotropism (ranging from imminent ovarian failure to full-blown POF), however, the better parameter to assess the extent of ovarian follicle depletion seems to be represented by AMH (Broekm 109). It is a dimeric glycoprotein with autocrine and paracrine actions in follicle development, exclusively produced by granulose cells of preantral (primary and secondary) and small antral follicles (2-7 mm in diameters). The number of small antral follicles is directly related to the total size of the primordial follicle pool (Broekm 68). With the decrease in the number of antral follicles with age, AMH serum levels also become diminished (Br 66, 95, 104) and will invariably become undetectable near menopause (Br 65). Recent studies have indeed suggested that AMH serum levels represent ovarian quantitative reserve (Br 105-107) and may provide an index of age at menopause.

Regarding ultrasound markers, several studies, recently, demonstrated that Antral Follicle Count (AFC), defined as the total number of antral follicles, sized 2-10 mm, present in both ovaries, represents a better marker than either chronological age or basal FSH for assessing the ovarian biological age [alviggi 89] and it has also been correlated with the occurrence of the menopausal transition (broekm 66), indicating that this parameter relates strongly with the quantitative aspects of ovarian reserve.

As for AFC, ovarian volume, measured by vaginal ultrasound, has been associated to the ovarian functional asset and also transvaginal ultrasound with the use of power Doppler is often used to evaluate the blood flow through the ovary in natural cycles. Several studies, moreover, have shown that ovarian flow index at the baseline ultrasound scan are correlated with subsequent follicular response and may be a new indicator for predicting ovarian responsiveness in IVF treatment (Sattar 2005) The added value of ovarian volume and stromal blood flow, however, either individually or together, to AFC and endocrine markers, in the predictability of ovarian age has not been assessed in a multivariate module.

The challenge of any ovarian reserve tests, anyhow, lies in the possibility of identifying women with a reduced reproductive life span at such an early stage in their lives that adequate action can be taken. Basal endocrine levels and sonographic parameters, however, are usually considered to have low specificity and sensitivity when used both to predict low ovarian reserve in infertile women (Younis 2010) and to prognosticate distance from menopause. Although these simple tests have been extensively investigated in the past they have seldom been looked into in combination. On the contrary, improvement of tests for the identification of women with a reduced ovarian life span will probably come from combining endocrine and imaging evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years
* Consent to participate to the prospective study
* Regular menses at 22 to 35 day interval

Exclusion Criteria:

* Estrogen or progestin-containing medications in the month before enrollment
* Gynecological malignancy
* Hypogonadotropic hypogonadism
* Assumption of drugs that can cause menstrual irregularity

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Ovarian Age prediction | One month
  Reliability of a multimodal diagnostic evaluation of ovarian age in term of both reproductive prognosis and distance to menopause

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, MD, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy

REFERENCES:
- [Result] Venturella R, Lico D, Sarica A, Falbo MP, Gulletta E, Morelli M, Zupi E, Cevenini G, Cannataro M, Zullo F. OvAge: a new methodology to quantify ovarian reserve combining clinical, biochemical and 3D-ultrasonographic parameters. J Ovarian Res. 2015 Apr 8;8:21. doi: 10.1186/s13048-015-0149-z. PMID 25881987
- [Result] Venturella R, Morelli M, Lico D, Di Cello A, Rocca M, Sacchinelli A, Mocciaro R, D'Alessandro P, Maiorana A, Gizzo S, Zullo F. Wide excision of soft tissues adjacent to the ovary and fallopian tube does not impair the ovarian reserve in women undergoing prophylactic bilateral salpingectomy: results from a randomized, controlled trial. Fertil Steril. 2015 Nov;104(5):1332-9. doi: 10.1016/j.fertnstert.2015.08.004. Epub 2015 Aug 31. PMID 26335129
- [Result] Venturella R, Lico D, Borelli M, Imbrogno MG, Cevenini G, Zupi E, Zullo F, Morelli M. 3 to 5 Years Later: Long-term Effects of Prophylactic Bilateral Salpingectomy on Ovarian Function. J Minim Invasive Gynecol. 2017 Jan 1;24(1):145-150. doi: 10.1016/j.jmig.2016.08.833. Epub 2016 Sep 13. PMID 27621194